CLINICAL TRIAL: NCT05725681
Title: The Role of High-Protein Instant Ramen Noodles in Inducing and Maintaining Satiety: Acute, Randomized, Crossover Study
Brief Title: Satiety of High-Protein Ramen Noodles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 22-0729
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein ramen (Experimental): Participants will be asked to limit physical activity to a specified level, consume a standardized meal at night and report to the clinic after a 12 h overnight fast. At our clinic, for this arm, participants will consume one portion of high-protein instant ramen noodles (71 g; Chef Woo, Borealis Foods). In the 4-hours following the ramen breakfast, blood will be sampled at regular intervals (0 minutes - before starting the breakfast, and 30, 60, 120 and 180 minutes after stopping breakfast) for hunger and satiety hormones (i.e., glucagon like peptide-1, peptide-YY, and ghrelin), and glucose and insulin. Visual Analogue Scales will also be administered to assess subjective hunger and satiety. At 4-hours, a buffet-style lunch will be provided and caloric intake at the meal will be covertly assessed.
  Interventions: Other: High protein ramen
- Standard ramen (Active Comparator): Participants will be asked to limit physical activity to a specified level, consume a standardized meal at night and report to the clinic after a 12 h overnight fast. At our clinic, for this arm, participants will consume an isocaloric, weight matched portion of standard instant ramen noodles. In the 4-hours following the ramen breakfast, blood will be sampled at regular intervals (0 minutes - before starting the breakfast, and 30, 60, 120 and 180 minutes after stopping breakfast) for hunger and satiety hormones (i.e., glucagon like peptide-1, peptide-YY, and ghrelin), and glucose and insulin. Visual Analogue Scales will also be administered to assess subjective hunger and satiety. At 4-hours, a buffet-style lunch will be provided and caloric intake at the meal will be covertly assessed.
  Interventions: Other: Standard ramen

INTERVENTIONS:
Other: High protein ramen — Participants will be served one portion of high-protein instant ramen noodles [CHEF WOO Roasted Chicken Flavor Ramen Cup Noodles, Borealis Foods; 71 g]
  Arms: High protein ramen
Other: Standard ramen — Participants will be served one portion of standard instant ramen noodles [RAMEN EXPRESS Chicken Flavor Ramen Cup Noodle Chef Woo, Borealis Foods; 71 g]
  Arms: Standard ramen

SUMMARY:
The aim of this study is to determine if high-protein instant ramen noodles acutely increase satiety, reduce hunger, and improve blood sugar levels compared to standard instant ramen noodles in generally healthy young to middle aged adults. In addition, investigators aim to test if intake of high-protein instant ramen noodles reduces caloric intake at the next meal compared to standard instant ramen noodles.

DETAILED DESCRIPTION:
The aim of this study is to determine if high-protein instant ramen noodles acutely increase satiety, reduce hunger, and improve blood sugar levels compared to standard instant ramen noodles in generally healthy young to middle aged adults. In addition, investigators aim to test if intake of high-protein instant ramen noodles reduces caloric intake at the next meal compared to standard instant ramen noodles. Subjects meeting the eligibility criteria will be recruited and offered a 2-condition, randomized, crossover postprandial study. Participants will be asked to limit physical activity to a specified level, consume a standardized meal at night and report to the clinic after a 12 h overnight fast. At our clinic, in random order, participants will consume: 1) one portion of high-protein instant ramen noodles (71 g; Chef Woo, Borealis Foods); 2) an isocaloric, weight matched portion of standard instant ramen noodles. The participants will have to finish consuming the noodles within 15 minutes. Water will be provided at the time of breakfast and for the next two hours. In the 4-hours following the ramen breakfast, blood will be sampled at regular intervals (0 minutes - before starting the breakfast, and 30, 60, 120 and 180 minutes after stopping breakfast) for hunger and satiety hormones (i.e., glucagon like peptide-1, peptide-YY, and ghrelin), and glucose and insulin. Visual Analogue Scales will also be administered to assess subjective hunger and satiety. At 4-hours, a buffet-style lunch will be provided and caloric intake at the meal will be covertly assessed. Subjects will leave the clinic at this point. The process will be repeated for the second condition after at least 7 d washout period.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index 20-30 kg/m2

Exclusion Criteria:

* Unwilling or unable to have an IV catheter inserted
* Body weight <110 pounds
* Diabetes (any type)
* Fasting capillary glucose ≥100 mg/dL
* Unstable systemic medical condition

  •>10% change in body weight in the prior 3 months
* Medications that affect appetite or glucose regulation
* Prior bariatric surgery
* Uncontrolled hypertension (i.e., unmedicated blood pressure >130/90 mmHg)
* Intolerance, dislike or allergy to the study food
* Current or recent (within 6 months) tobacco use
* High alcohol consumption (>14 drinks/week)
* Currently following a weight loss diet
* Irregular menstrual cycle
* Currently pregnant or lactating
* Principal investigator discretion (e.g., disrespectful or inappropriate interactions with study staff

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Appetite Score Area Under the Curve (mm*180 minutes) | 0 to 180 minutes
  Calculated as satiety + fullness + (100 - hunger) + (100 - prospective food consumption)/4. Questions 1-4 from the Visual Analogue Scale will be used to assess satiety, fullness, hunger and prospective food consumption and calculate the Appetite Score

SECONDARY OUTCOMES:
Ghrelin Area Under the Curve (pg/mL*180 minutes) | 0 to 180 minutes
  Measured in plasma
Glucagon like peptide-1 (GLP-1) Area Under the Curve (pg/mL*180 minutes) | 0 to 180 minutes
  Measured in plasma
Peptide-YY (PYY) Area Under the Curve (pg/mL*180 minutes) | 0 to 180 minutes
  Measured in plasma
Glucose Area Under the Curve (mg/dL*180 minutes) | 0 to 180 minutes
  Measured in plasma
Insulin Area Under the Curve (mUI*180 minutes) | 0 to 180 minutes
  Measured in serum
Perceived Hunger Area Under the Curve (mm*180 minutes) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived Satiety Area Under the Curve (mm*180 minutes) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived Fullness Area Under the Curve (mm*180 minutes) | 0 to 180 minutes
  Assessed by visual analogue scale.
Prospective Food Consumption Area Under the Curve (mm*180 minutes) | 0 to 180 minutes
  Assessed by visual analogue scale.
Minimum ghrelin (pg/mL) | 0 to 180 minutes
  Measured in plasma
Peak Glucagon like peptide-1 (GLP-1) (pg/mL) | 0 to 180 minutes
  Measured in plasma
Peak Peptide-YY (PYY) (pg/mL) | 0 to 180 minutes
  Measured in plasma
Peak Glucose (mg/dL) | 0 to 180 minutes
  Measured in plasma
Peak Insulin (mUI) | 0 to 180 minutes
  Measured in serum
Desire to eat something fatty Area Under the Curve (mm*180 minutes) | 0 to 180 minutes
  Assessed by visual analogue scale.
Desire to eat something salty Area Under the Curve (mm*180 minutes) | 0 to 180 minutes
  Assessed by visual analogue scale.
Desire to eat something savory Area Under the Curve (mm*180 minutes) | 0 to 180 minutes
  Assessed by visual analogue scale.
Desire to eat something sweet Area Under the Curve (mm*180 minutes) | 0 to 180 minutes
  Assessed by visual analogue scale.
Energy intake at the buffet lunch (kcal) | Served approximately 3.5 hours following the ramen meal test
  Food consumed during the buffet lunch
Perceived hunger at peak GLP1 (mm) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived satiety at peak GLP1 (mm) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived fullness at peak GLP1 (mm) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived hunger at peak PYY (mm) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived satiety at peak PYY (mm) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived fullness at peak PYY (mm) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived hunger at minimum ghrelin (mm) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived satiety at minimum ghrelin (mm) | 0 to 180 minutes
  Assessed by visual analogue scale.
Perceived fullness at minimum ghrelin (mm) | 0 to 180 minutes
  Assessed by visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Dhurandhar, Principal Investigator — Department of Nutritional Sciences Texas Tech University; Kristina Petersen, Principal Investigator — Department of Nutritional Sciences Texas Tech University
Locations (1):
- Nutrition and Metabolic Health Initiative, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code